# Q-Med AB, part of the Galderma Group

A Prospective, Non-interventional Study to Collect Subject and Physician Satisfaction During Long Term Treatment of Glabellar Lines with Dysport® in Subjects of Chinese Origin in Real Clinical Practice

05PF2009

Statistical Analysis Plan

Version: 2.0

Date: 15Mar2024

# APPROVAL PAGE

A Prospective, Non-interventional Study to Collect Subject and Physician Satisfaction During Long Term Treatment of Glabellar Lines with Dysport® in Subjects of Chinese Origin in Real Clinical Practice

# 05PF2009

# Statistical Analysis Plan Version: 2.0

| Prepared by | y: | |
|-------------|-----|------|
| PPD | | |
| Reviewed 1 | by: | |
| Approved 1 | by: | <br> |
| PPD | | |

# MODIFICATION HISTORY

| VERSION | VERSION DATE | AUTHOR | DESCRIPTION |
|---|---|---|---|
| 1.0 | 2024.02.19 | PPD | FINAL VERSION |
| 2.0 | 2024.03.15 | | All adverse reactions were revised to adverse events; |
| | | | TFL is updated according to the ICH-E3 standard |

# **TABLE OF CONTENTS**

| Al | BBREV | TATION | 6 |
|----|--------|-------------------------------------|-----|
| 1. | INT | RODUCTION | 7 |
| 2. | STU | JDY OBJECTIVE | 7 |
| 3. | STU | UDY DESIGN | 7 |
| | 3.1. | Investigational Product (IP) | 7 |
| | 3.2. | Study Flow Chart | 7 |
| | 3.3. | Schedule of Assessments | 8 |
| | 3.4. | Randomization Design and Execution | 8 |
| | 3.5. | Blinding Design and Execution. | 8 |
| | 3.6. | Sample Size Consideration. | 8 |
| 4. | EN | DPOINTS | 8 |
| | 4.1. | Efficacy Endpoints | 8 |
| | 4.2. | Safety Endpoints | 9 |
| | 4.3. | Demographics and Disease Characters | 0 |
| | 4.4. | Prior/Concomitant Medication | 0 |
| | 4.5. | Prior/Concomitant Treatment | 1 |
| | 4.6. | Protocol Deviation | 1 |
| 5. | STA | ATISTICAL HYPOTHESIS1 | . 1 |
| 6. | AN | ALYSIS SETS1 | . 1 |
| | 6.1. | Full Analysis Set (FAS) | 1 |
| | 6.2. | Per Protocol Set (PPS) | 1 |
| | 6.3. | Safety Set (SS) | 1 |
| 7. | STA | ATISITICAL METHODS1 | . 1 |
| | 7.1. | General Statistical Consideration | 1 |
| | 7.1.1. | Application of Analysis Sets1 | .1 |
| | 7.1.2. | Descriptive Statistics | .1 |
| | 7.1.3. | Decimals1 | 2 |
| | 7.1.4. | General Statistical Test Methods1 | 2 |
| | 715 | Significance Level | 2 |

| 7.1.6. | Software for Statistical Analysis | 2 |
|--------|--------------------------------------------|---|
| 7.1.7. | Definition of Baseline1 | 2 |
| 7.1.8. | Scheduled and Unscheduled Visit | 3 |
| 7.1.9. | Subject Identifier 1 | 3 |
| 7.2. | Data Handling1 | 3 |
| 7.3. | Subjects in Study1 | 3 |
| 7.3.1. | Subjects Disposition1 | 3 |
| 7.3.2. | Protocol Deviation1 | 3 |
| 7.3.3. | Analysis Sets | 3 |
| 7.3.4. | Demographics and Baseline Characters 1 | 4 |
| 7.3.5. | Allergy History1 | 4 |
| 7.3.6. | Prior/Concomitant Medication1 | 4 |
| 7.3.7. | Prior/Concomitant Treatment1 | 4 |
| 7.4. | Efficacy Analysis1 | 5 |
| 7.4.1. | Analysis on Primary Efficacy Endpoints 1 | 5 |
| 7.4.2. | Analysis on Secondary Efficacy Endpoints 1 | 5 |
| 7.5. | Safety Analysis1 | 5 |
| 7.6. | Interim Analyses | 6 |
| 7.7. | Change from the Analysis Plan in Protocol | 6 |
| 8. REF | ERENCE1 | 7 |
| 9. TFL | SHELL | 7 |

# **ABBREVIATION**

| Abbreviation | Specification |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| AE | Adverse Event |
| ATC | Anatomical Therapeutic Chemical |
| BoNT | Botulinum toxin |
| BoNT-A | Botulinum toxin serotype A |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| GCP | Good Clinical Practice |
| GL | Glabellar lines |
| FAS | Full Analysis Set |
| ICH | International Council for Harmonization |
| IP | Investigational Product |
| MedDRA | Medical Dictionary For Regulatory Activities |
| NA | Not Applicable |
| NMPA | National Medical Products Administration |
| PPS | Per Protocol Set |
| PT | Preferred Term |
| Q1 | 25% quartile |
| Q3 | 75% quartile |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAR | Statistical Analysis Report |
| SAS | Statistical Application Software |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Events |
| SS | Safety Set |
| SS Event | Special Situation Event |
| UAE | Unexpected Adverse Drug Reaction |
| WHO DD | World Health Organization Drug Dictionary |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the statistical methods that will be used in summarizing and analyzing the efficacy and safety data that will be collected in this study 05PF2009 and aims to support the clinical study report (CSR). This statistical analysis plan will be finalized prior to database lock.

This document is developed based on the protocol version 2.0 (28 Jun 2021) and electronic Case Report Form (eCRF) version 1.1 (01 Jan2023) and compliances with the recommendations of the International Conference on Harmonization (ICH) E9 guidelines "Statistical Principles for Clinical Trials" [1] and the ICH E3 guidelines "Structure and Content of Clinical Study Reports" [2].

## 2. STUDY OBJECTIVE

To collect subject and physician satisfaction, and treatment experience with Dysport in real clinical practice in subjects of Chinese origin.

#### 3. STUDY DESIGN

This is a prospective, longitudinal, non-interventional, multi-center study.

### 3.1.Investigational Product (IP)

Commercially available Dysport, a BoNT-A product, strength: 300U per vial, produced and supplied by Q-Med AB, part of the Galderma Group.

### 3.2.Study Flow Chart

Study Flow Chart is shown below.



#### 3.3. Schedule of Assessments

Schedule of Assessments of the study is shown below.

| | Injection Cycle 1 | | Injection Cycle 2 | | Injection Cycle 3 | | |
|---|---|---|---|---|---|---|---|
| Visit Number | Visit 1 <sup>1</sup> | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
| Visit Name | Screening<br>Baseline/Injection 1 <sup>1</sup> | Follow up 1 | Injection 2 | Follow up 2 | Injection 3 | Follow up 3 | Follow up 4 |
| Visit Window | ≤ 30 days of<br>Baseline/Injection 1 | 3 weeks (± 7 days)<br>from Injection 1 | 3-6 months<br>from Injection 1 | 3 weeks (± 7 days)<br>from Injection 2 | 3-6 months<br>from Injection 2 | 3 weeks (± 7 days)<br>from Injection 3 | 3-6 months<br>from Injection 3 |
| Informed Consent | X | | | | | | |
| Demographic Data | X | | | | | | |
| Medical History | X | | | | | | |
| Safety Review | X | X | X | X | X | X | X |
| Injection Practice Details | X | | X | | X | | |
| Physician GL Severity Assessment | X <sup>2</sup> | X | X <sup>2</sup> | X | $X^2$ | X | X |
| Physician Satisfaction Questionnaire | X <sup>2</sup> | X | $X^2$ | X | $X^2$ | X | X |
| Subject assessments | | | | | | , | |
| Subject GL Severity Assessment | X <sup>2</sup> | X | X <sup>2</sup> | X | $X^2$ | X | X |
| Subject Satisfaction Questionnaire | X <sup>2</sup> | X | X <sup>2</sup> | X | X <sup>2</sup> | X | X |

 <sup>1</sup> month = 4 weeks

### 3.4. Randomization Design and Execution

Not applicable. This is a non-interventional study.

### 3.5.Blinding Design and Execution

Not applicable. This is a non-interventional study.

### 3.6. Sample Size Consideration

The sample size of approximately 250 subjects is not based on a statistical calculation. The selected number of subjects is regarded as sufficient for an evaluation of the studied endpoints by using descriptive statistics.

#### 4. ENDPOINTS

## 4.1. Efficacy Endpoints

### 4.1.1. Primary Efficacy Endpoints

The primary efficacy endpoint is subject satisfaction after three injection cycles with Dysport with GL. At Visit 6 subjects will be asked "What is your overall satisfaction after three treatments cycles with Dysport?" Response options are: very satisfied, satisfied, dissatisfied, and very dissatisfied. The primary endpoint will evaluate the proportion of subjects in each response category.

### 4.1.2. Secondary Efficacy Variables

<sup>1.</sup> Screening and Baseline/Visit 1 (i.e., Injection 1) may be performed on the same day. If performed as separate visits, informed consent, demographic data, and medical history should be complete at Screening, and all other remaining visit procedures and confirmation of subject medical history should be performed at Baseline/Visit 1 (i.e., Injection 1).

<sup>2.</sup> Prior to injection.

1 Physician satisfaction after three injection cycles with Dysport in the GL. The proportion of subjects in each response category for the physician's overall satisfaction with Dysport at Visit 6.

② a. Proportions of subjects in each response category per question answered on the Subject Satisfaction Ouestionnaire complete at all visits.



# **4.2.Safety Endpoints**

### 4.2.1. Adverse Event (AE)

Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory

finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.

Thus, any new sign, symptom or disease, or any clinically significant worsening of an existing sign, symptom or disease (including new episodes of a chronic disease) compared to the condition at the first visit, should be considered as an AE.

### 4.2.2. Unexpected Adverse Event (UAE)

An unexpected AE is defined as an adverse event, the nature or severity of which is not consistent with the applicable study product information (e.g., medicinal package insert/summary of product characteristics for an approved study product).

### 4.2.3. Serious Adverse Event (SAE)

A SAE is any untoward medical occurrence that at any dose:

- (1) Results in death
- (2) Is life-threatening
- (3) Requires inpatient hospitalization or prolongation of existing hospitalization
- (4) Results in persistent or significant disability/incapacity
- (5) Is a congenital anomaly/birth defect

### 4.2.4. Special Situation (SS) Events

SS Event is an incidence of overdose, off-label use, medication error, occupational exposure, abuse, misuse, or lack of therapeutic efficacy while using the medicinal product, or any instance of drug exposure during pregnancy or breast-feeding.

### 4.2.5. Severity

- (1) Mild: Awareness of signs or symptom, but easily tolerated.
- (2) Moderate: Discomfort, enough to cause interference with usual activity.
- (3) Severe: Incapacitating with inability to work or perform usual activity.

# 4.3. Demographics and Disease Characters

#### 4.3.1. Demographics

The demographics including age, sex, and nation will be recorded in CRF.

### 4.3.2. Medical History

The information of medical history including disease name, start date, end date and ongoing will be recorded in CRF.

## 4.3.3. Surgery History

The name and date of surgery prior to screening will be recorded in CRF.

### 4.3.4. Allergy History

The information of allergy history will be recorded in CRF.

#### 4.4. Prior/Concomitant Medication

The information of prior/concomitant medication including drug name, dose, unit, frequency, route of administration, start date, end date, ongoing, and reason for usage will be recorded in CRF.

#### 4.5. Prior/Concomitant Treatment

The information of prior/concomitant treatment including name of treatment, start date, end date, ongoing, and treatment reason will be recorded in CRF during the study.

#### 4.6.Protocol Deviation

Clinical operation team shall record the cause, date and severity of all protocol deviations in the file Protocol Deviation Tracking Log.

### 5. STATISTICAL HYPOTHESIS

Not applicable. This is a non-interventional study.

### 6. ANALYSIS SETS

### **6.1.Full Analysis Set (FAS)**

All subjects screened, enrolled in the study treated at least once with Dysport.

### **6.2.Per Protocol Set (PPS)**

A subset of FAS that include subjects who have evaluable primary efficacy endpoints, have overall good compliance, and have no major protocol deviations during the study. Subjects excluded from PPS will be determined in Data Review Meeting before Data Base Lock.

## 6.3. Safety Set (SS)

The set of subjects who have received at least one dose of study treatment and for whom actual data on safety endpoints are available.

#### 7. STATISITICAL METHODS

#### 7.1. General Statistical Consideration

Demographics and disease characteristics data, efficacy data, and safety data will be analyzed. The annotated or explanatory transcript will only be listed. The following rules apply to general situations unless otherwise stated.

#### **7.1.1.** Application of Analysis Sets

Baseline analyses will be based on FAS and PPS; efficacy analyses will be primarily based on PPS, and on FAS as reference; safety analyses will be based on SS.

#### **7.1.2.** Descriptive Statistics

For continuous data, descriptive statistics include number of non-missing patients, number of missing patients (nmiss), mean, standard deviation (SD), median, Q1, Q3, minimum, and maximum.

Statistical Analysis Plan Version: 2.0

For categorical data, the frequency and percentage of patients in each category will be presented. Counts that are zero will be displayed as "0". Percentages will be based on non-missing data unless otherwise specified. Two-sided 95% confidence interval will be calculated for the estimated incidence wherever appropriate.

#### 7.1.3. Decimals

The minimum and maximum will keep the same decimal place with the raw data, while mean, median, Q1 and Q3 will keep 1 more decimal place, and SD will keep 2 more decimal places. The decimal place of above statistics will not exceed 4 regardless of the decimal place of raw data.

Percentages and 95% confidence interval (CI) will keep 1 decimal place.

P value will be rounded to 4 decimal places. '<.0001' will be displayed when the P value is lesser than 0.0001 and '>.9999' will be displayed when the P value is greater than 0.9999.

#### **7.1.4.** General Statistical Test Methods

For continuous data, parametric or non-parametric method will be used according to the result of Shapiro-Wilk test with 5% significance level.

For within-group comparison, paired t-test will be performed if the assumption of normality is satisfied, otherwise Wilcoxon signed rank test will be performed.

For between-group comparison, two sample t-test will be performed if the assumption of normality is satisfied, otherwise Wilcoxon rank sum test will be performed.

For between-group comparison of categorical data, chi-square test will be basically performed and the Wald asymptotic 95% confidence interval will be calculated.

But in case of more than 20% of the number of cells with an expected frequency of less than 5, Fisher's exact test will be performed and the exact 95% confidence intervals will be calculated.

### **7.1.5.** Significance Level

Statistical analysis will be performed with a two-sided test at a significance level of 5% whenever required.

#### **7.1.6.** Software for Statistical Analysis

Statistical programming will use SAS® 9.4 or higher version.

### 7.1.7. Definition of Baseline

The baseline values for all variables (if applicable) are defined as the latest measurement or examine result before injection.

#### 7.1.8. Scheduled and Unscheduled Visit

Generally, statistical description by visits will be performed on the scheduled visits unless it is specified otherwise. For shift table of clinical evaluation of safety data, the data on scheduled and unscheduled visits will be all included in the analyses.

### **7.1.9.** Subject Identifier

For the data listing, screening number (USUBJID) will be used as a unique identifier.

## 7.2.Data Handling

Data will be analyzed as observed without imputation for missing values.

### 7.3. Subjects in Study

### 7.3.1. Subjects Disposition

The following summaries will be tabulated:

- No. and percentage of subjects screened and reasons for screening failure
- No. and percentage of subjects who are treated and not treated.
- No. and percentage of subjects who completed the study.
- No. and percentage of subjects who prematurely discontinued study and reasons of early termination

The above analysis will be summarized for each site.

Detailed information regarding disposition of each subject will be listed.

#### 7.3.2. Protocol Deviation

For all enrolled subjects, all major protocol deviations recorded by clinical operation team will be summarized according to predefined categories. All the protocol deviations will be recorded in the file Protocol Deviation Tracking Log.

Major protocol deviations will be summarized for each site.

All protocol deviations recorded by clinical operation team of each subject will be listed.

## **7.3.3.** Analysis Sets

For all enrolled subjects, the number of subjects in each analysis set will be summarized together with the number of subjects excluded from each analysis set and the corresponding reasons.

The above analysis will be summarized for each site.

Detailed information of analysis sets will be listed.

### **7.3.4.** Demographics and Baseline Characters

# Demographics

The demographics including age, sex, and nation will be summarized using descriptive statistics.

Detailed information of demographics will be listed by subject.

### Medical/ Surgery History

Number of events, number and percentage of subjects who had at least one medical history will be summarized using descriptive statistics. All medical history will also be summarized by System Organ Class (SOC) and preferred term (PT) that will be coded using the MedDRA version 25.1.

Detailed information of medical/surgery history will be listed by subject.

### **7.3.5.** Allergy History

Number of events, number and percentage of subjects who had at least one allergy history will be summarized using descriptive statistics. The number of events will also be presented.

Detailed information of allergy history will be listed by subject.

#### **7.3.6.** Prior/Concomitant Medication

Prior medication and concomitant medication analyses will be based on FAS and PPS.

Prior medication and concomitant medications will be coded by the World Health Organization Drug Dictionary (WHO DD) Global (B3) E [V2022SEP]. Prior and concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) classification (including Anatomy group, Therapeutic group and Chemical group) and WHO preferred drug name, respectively. The summary will be sorted in decreasing order of percentage of ATC class firstly and then sorted in decreasing order of percentage of preferred drug term within the ATC class.

Prior medications: if the end date of the medication is before the date of injection in this study. Concomitant medications: if the end date of the medication is on or after the date of injection in this study or still ongoing.

Detailed information of prior and concomitant medications will be listed by subject.

#### **7.3.7.** Prior/Concomitant Treatment

Prior and concomitant treatment analyses will be based on FAS and PPS.

Number of events, number and percentage of subjects who had at least one treatment will be summarized using descriptive statistics.

All prior/concomitant treatment will be coded by MedDRA version 25.1 and summarized by SOC and PT.

Detailed information of prior/concomitant treatment will be listed by subject.

# 7.4. Efficacy Analysis

## **7.4.1.** Analysis on Primary Efficacy Endpoints

Analysis on primary efficacy endpoints will be performed on PPS and FAS.

At Visit 6 proportion of subjects in each response category from subject satisfaction will be evaluated and its exact 95% CI will be calculated.

# **7.4.2.** Analysis on Secondary Efficacy Endpoints

Analysis on secondary efficacy endpoints will be performed on PPS and FAS.

- ① At Visit 6 proportion of subjects in each response category from physician overall satisfaction will be evaluated and its exact 95% CI will be calculated.
- ② a. At all visits proportion of subjects in each response category per question from subject satisfaction will be evaluated and its exact 95% CI will be calculated.



### 7.5. Safety Analysis

AEs will be coded by MedDRA version 25.1. SOC and PT will be presented in summary tables of AE. All summary table will be based on Treatment Emergent AE (TEAE).

TEAE defines as all AEs that occur after the first treatment.

Overall TEAEs, UAEs, SAEs, SS Events, AEs leading to discontinuation from study, AEs leading to death and whether these AEs are possibly caused by the product and/or injection procedure, will be summarized by number of events, number of subjects, percentage and 95% CI.

The number of events, number of subjects and percentage with AEs and product and/or injection procedure related AEs will be summarized for each category by SOC, PT and severity. If multiple

AEs in the same SOC (PT) have occurred in the same subject when summarizing the number of subjects, the subject will be counted only once for this SOC (PT). When summarizing the number of subjects by severity, if multiple AEs in the same SOC (PT) have occurred in the same subject, the event with the highest severity of this SOC (PT) will be used for analysis. When summarizing the number of events, all the AEs will be accounted.

Detailed information of AEs, UAEs, SAEs, SS Events, AEs possibly caused by the product and/or injection procedure, AEs leading to discontinuation, and AEs leading to death will be listed by subject.

# 7.6.Interim Analyses

Two interim analyses will be performed before the final analysis. The first interim analysis will be performed after Visit 2. The second interim analysis will be performed after Visit 4. Only applicable tables and listings will be generated for interim analyses.

### 7.7. Change from the Analysis Plan in Protocol

Two interim analyses are added after the first two injection cycles before the final analysis.

| Section | Description in protocol | Description in SAP |
|---|---|---|
| 4.2.1 | Adverse Drug Reaction (ADR) For marketed medicinal products, an ADR is a response to a drug which is noxious and unintended and which occurs at doses normally used in man for prophylaxis, diagnosis, or therapy of diseases or for modifications of physiological function. | delete |
| 4.2.2 | Unexpected Adverse Drug Reaction (UADR) An unexpected ADR is defined as an adverse reaction, the nature or severity of which is not consistent with the applicable study product information (e.g.,medicinal packageinsert/summary of product characteristics for an approved study product). | Unexpected Adverse Event (UAE) An unexpected AE is defined as an adverse event, the nature or severity of which is not consistent with the applicable study product information (e.g., medicinal package insert/summary of product characteristics for an approved study product). |

# 8. REFERENCE

- [1] ICH E9: Statistical Principles for Clinical Trials (1998).
- [2] ICH E3: Structure and Content of Clinical Study Reports (1995).

# 9. TFL SHELL

Refer to the attached document of SAP.



| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 3/18/2024 6:03:48 PM |
| Certified Delivered | Security Checked | 3/19/2024 10:06:29 AM |
| Signing Complete | Security Checked | 3/19/2024 10:06:42 AM |
| Completed | Security Checked | 3/19/2024 10:06:42 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, SoftwareOne OBO Galderma International (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact SoftwareOne OBO Galderma International:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: docusign support@galderma.com

### To advise SoftwareOne OBO Galderma International of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at docusign\_support@galderma.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from SoftwareOne OBO Galderma International

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to docusign\_support@galderma.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with SoftwareOne OBO Galderma International

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to docusign\_support@galderma.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify SoftwareOne OBO Galderma International as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by SoftwareOne OBO Galderma International during the course of your relationship with SoftwareOne OBO Galderma International.